CLINICAL TRIAL: NCT01529957
Title: A Phase I Clinical Study of Nemonoxacin Malate Sodium Chloride Injection Administered by Intravenous Infusion
Brief Title: A Study of Nemonoxacin Malate Sodium Chloride Injection Administered by Intravenous Infusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG-873870-C-2
Record Dates: First submitted 2012-02-03; First posted 2012-02-09 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Nemonoxacin Malate Sodium Chloride 25 mg (Active Comparator): Nemonoxacin Malate Sodium Chloride 25 mg
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride
- Nemonoxacin Malate Sodium Chloride 50 mg (Active Comparator): Nemonoxacin Malate Sodium Chloride 50 mg
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride
- Nemonoxacin Malate Sodium Chloride 125 mg (Active Comparator): Nemonoxacin Malate Sodium Chloride 125 mg
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride
- placebol (Placebo Comparator): placebol
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride
- Nemonoxacin Malate Sodium Chloride 250 mg (Active Comparator): Nemonoxacin Malate Sodium Chloride 250 mg
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride
- Nemonoxacin Malate Sodium Chloride 500 mg (Active Comparator): Nemonoxacin Malate Sodium Chloride 500 mg
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride
- Nemonoxacin Malate Sodium Chloride 650 mg (Active Comparator): Nemonoxacin Malate Sodium Chloride 650 mg
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride
- Nemonoxacin Malate Sodium Chloride 750 mg (Active Comparator): Nemonoxacin Malate Sodium Chloride 750 mg
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride
- Nemonoxacin Malate Sodium Chloride 1000 mg (Active Comparator): Nemonoxacin Malate Sodium Chloride 1000 mg
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride
- Nemonoxacin Malate Sodium Chloride 1250 mg (Active Comparator): Nemonoxacin Malate Sodium Chloride 1250 mg
  Interventions: Drug: Nemonoxacin Malate Sodium Chloride

INTERVENTIONS:
Drug: Nemonoxacin Malate Sodium Chloride — Nemonoxacin Malate Sodium Chloride,intravenous injection,once daily

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of nemonoxacin in healthy Chinese volunteers.

DETAILED DESCRIPTION:
Single dose safety and tolerability study: evaluate safety and tolerability of intravenous infusion nemonoxacin 25mg, 50mg, 125mg, 250mg, 500mg, 750mg, 1000mg and 1250mg.

Single dose pharmacokinetic (PK) study:evaluate PK profile of doses of 250mg, 500mg or 750mg intravenous infusion nemonoxacin .

Multiple dose study: evaluate PK profile of doses of 500mg, 650mg or 750mg intravenous infusion nemonoxacin after consecutive 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, aged 18 ~45
2. A male volunteer should be willing to use a double-barrier contraception until the study is completed, and should not make his partner pregnant during the study and within 3 months after completing the study
3. Volunteers who have never used any tobacco or nicotine-containing product within three months before use of the investigational product
4. Volunteers who are willing to abstain from caffeine- or xanthine- containing drinks or food within 24h before being enrolled in the study and throughout the study,such as coffee and tea,chocolate,alcohol, grapefruit juice,orange juice,etc.
5. The body mass index (BMI) of the volunteer must be 19~24, and the weight of a male should be at least 50kg,and that of a female should be at least 45kg.
6. Volunteers who are able to sign the informed consent form (ICF) of their own accord.

Exclusion Criteria:

1. History of diabetes,or cardiovascular,hepatic or renal disease.
2. Had surgery or trauma within 6 months prior to this study
3. Alcohol or drug abuse
4. HIV, HBV or HCV positive
5. subject used any known hepatic enzyme inducer/hepatic enzyme inhibitor product within 30 days prior to the study
6. Used any prescribed drug (including traditional chinese medicine) within 14 days prior to the study
7. Donated 400ml of blood or plasma within 3 months prior to this study
8. Have an abnormal laboratory examination value that exceeds the normal range by 10%
9. Drug allergies
10. Have cardiac disorders or have a family history of cardiac disorders
11. Have abnormal 12-lead ECG during screening
12. Pregnant or lactating
13. Participated in any study within 3 months prior to this study
14. according to the investigator's judgment, affect the safety or efficacy evaluation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Adverse event assessment in healthy Chinese volunteer | 46days
Maximum tolerated single dose of nemonoxacin in healthy Chinese volunteers | 32days

SECONDARY OUTCOMES:
Pharmacokinetic profile of nemonoxacin in healthy Chinese volunteers | 4days

CONTACTS AND LOCATIONS:
Overall Officials: Yingyuan Zhang, PhD, Principal Investigator — Huashan Hospital, Fundan University
Locations (26):
- China (26):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Zhen Hospital, Capital Medical University Beijing, Beijing
  - Kunming General Hospital of Chengdu Military Region, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Second Affiliated Hospital, Third Military Medical University, Chongqing
  - Third Military Medical University First Affiliated Hospital, Chongqing
  - Third Military Medical University, Third Affiliated Hospital, Chongqing
  - Second Affiliated Hospital of Dalian Medical University, Dalian
  - Gansu Provincial People's Hospital, Gansu
  - Guangzhou Red Cross Hospital, Guangzhou
  - Second Affiliated Hospital of Sun Yat-sen, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - Third Xiangya Hospital, Central South University, Hunan
  - Xiangya Hospital, Central South University, Hunan
  - Jiangxi Provincial People's Hospital, Jiangxi
  - Second Affiliated Hospital of Nanchang University, Jiangxi
  - Shengjing Hospital of China Medical University, Liaoning
  - Huai'an First Hospital of Nanjing Medical University, Nanjing
  - Affiliated Hospital of Qingdao University Medical College, Qingdao
  - Institute of Antibiotics, Huashan Hospital, Fundan University, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai Pudong New Area, Oriental Hospital, Shanghai
  - People's Liberation Army General Hospital of Shenyang Military Region, Shenyang
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - First Affiliated Hospital,Zhejiang University School of Medicine, Zhejiang